CLINICAL TRIAL: NCT00839150
Title: Assessment of Retinal Functional Abnormalities in Diabetic Patients Without Retinopathy
Brief Title: Retinal Function in Diabetic Patients Without Retinopathy
Acronym: NEURODIAB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P041009
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetic retinopathy; Color vision; Contrast sensitivity; Electroretinogram; Flicker-induced vasodilatation; Dynamic Vessel Analyzer
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Diabetic patients without diabetic retinopathy : No intervention
- 2: Sex and age-matched control subjects : No intervention

SUMMARY:
The primary purpose was to assess, in diabetic patients without diabetic retinopathy and control subjects, color vision, contrast sensitivity, electroretinography, and flicker-induced vasodilatation using the Dynamic Vessel Analyzer, in order to specify the earliest impaired retinal cells in diabetes, and gain more insight into diabetic retinopathy pathogenesis.

DETAILED DESCRIPTION:
Type 1 and type 2 diabetic patients with no diabetic retinopathy and no hypertension were compared with sex and age-matched control subjects. Color vision was tested with the desaturated LANTHONY 15-Hue test. Contrast sensitivity was assessed with the Pelli-Robson contrast sensitivity test. Pattern-electroretinogram, Ganzfeld full-field electroretinogram and multifocal electroretinogram were recorded according to the International Society for Clinical Electrophysiology of Vision (ISCEV). Flicker-induced vasodilatation in retinal arteries and veins was assessed using the Dynamic Vessel Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* For diabetic patients :

  * age between 20 and 55
  * type 1 or type 2 diabetes mellitus
  * diabetes duration of more than 5 years
  * no diabetic retinopathy on fundus examination or fundus photographs
* For control subjects :

  * sex and age matching with the diabetic patients
  * no diabetes, no familial or personal history of elevated blood sugar

Exclusion Criteria:

*For both diabetic patients and control subjects :

* presence of cataract or history of cataract surgery
* intraocular pressure of more than 21 mmHg
* abnormal score on the Ishihara test
* other ocular disease
* ametropia more than 3 diopters, anisometropia more than 1 diopter, astigmatism more than 1 diopter
* systemic hypertension (defined as systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
* treatment with vasoactive drugs
* tobacco consumption of more than 20 cigarettes a day

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For diabetic patients :
  age between 20 and 55 type 1 or type 2 diabetes mellitus diabetes duration of more than 5 years no diabetic retinopathy on fundus examination or fundus photographs
  For control subjects :
  sex and age matching with the diabetic patients no diabetes, no familial or personal history of elevated blood sugar
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Massin, MD,Pr;PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Lariboisiere, Paris, France

REFERENCES:
- [Derived] Lecleire-Collet A, Audo I, Aout M, Girmens JF, Sofroni R, Erginay A, Le Gargasson JF, Mohand-Said S, Meas T, Guillausseau PJ, Vicaut E, Paques M, Massin P. Evaluation of retinal function and flicker light-induced retinal vascular response in normotensive patients with diabetes without retinopathy. Invest Ophthalmol Vis Sci. 2011 May 2;52(6):2861-7. doi: 10.1167/iovs.10-5960. PMID 21282578